CLINICAL TRIAL: NCT01942928
Title: Cranial Osteopathic Manipulative Therapy in Addition to Usual Care in Excessively Crying Infants, Sometimes Called Colic
Brief Title: Cranial Osteopathy in Infantile Colic
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: European School of Osteopathy (Other)
Collaborators: Sutherland Cranial College of Osteopathy (Unknown); Sutherland Society (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ESO-001-colic; ESO-001-2013 (Other: Sutherland Cranial College of Osteopathy)
Record Dates: First submitted 2013-09-11; First posted 2013-09-16 (Estimated); Last update posted 2015-02-20 (Estimated); Status verified 2015-02

CONDITIONS: Infantile Colic
MeSH Terms: conditions — Colic | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual NHS care (Active Comparator)
  Interventions: Other: Usual NHS Care
- Usual NHS Care plus Osteopathic Manipulative Therapy (Active Comparator)
  Interventions: Other: Usual NHS Care; Other: Osteopathic Manipulative Therapy

INTERVENTIONS:
Other: Usual NHS Care — Usual NHS care is provided by a health visitor who will diagnose excessively crying infants/infants with colic in the first instance. Parents usually will then have the opportunity to consult their health visitor when needed. The health visitor will provide support and advice on how to manage the condition within their professional remit.
Other: Osteopathic Manipulative Therapy — Osteopathic treatment will be provided by experienced osteopaths once a week for up to four weeks, depending on needs. Treatment will be individualised, according to clinical findings, and involves using standard cranial osteopathic techniques. All parents will be able to ask questions.
  Arms: Usual NHS Care plus Osteopathic Manipulative Therapy

SUMMARY:
Background Excessive Crying (Infantile Colic) is one of the most common complaints for which parents seek treatment. These otherwise healthy and well fed infants show no signs of failure to thrive, cry without identifiable cause, fuss a lot and are hard-to-soothe.

Objective To explore the feasibility of running a Randomised Controlled Trial (RCT) that investigates the effectiveness of cranial osteopathy in addition to usual National Health Service (NHS) care in infants with colic.

Methods Pragmatic randomised controlled trial, involving United Kingdom (UK) osteopaths in private practice and NHS health visitors. Parents of 60 excessively crying infants/infants with colic will be recruited by NHS health visitors. Infants will be included into the study if they are healthy (full-term) and aged 1-7 weeks, diagnosed with excessive crying/infantile colic, and have no co-morbidities. Participants will be randomised into the usual NHS care group or the usual NHS care plus cranial osteopathic intervention group.

Usual NHS care will be provided by health visitors and osteopathic treatment will be carried out by experienced osteopaths in private practice.

Primary outcome measures are acceptability and feasibility of intervention procedures. Furthermore, changes in the frequency and duration of crying will be documented in a daily crying diary. Parental quality of life will also be assessed.

This pilot investigation will provide useful information in order to further develop and adapt the current interventions and trial procedures with a view to a full-scale randomised controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* healthy, diagnosed with excessive crying by NHS Health Visitors No comorbidities Parents are able to adequately communicate in English

Exclusion Criteria:

* Currently participating in other therapeutic clinical trials Currently receive manual therapy treatment

Ages: 1 Week to 7 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change in daily hours crying time | 4 weeks

SECONDARY OUTCOMES:
Parental Quality of life | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- European School of Osteopathy, Maidstone, Kent, United Kingdom